CLINICAL TRIAL: NCT00778375
Title: Clofarabine Plus Low-Dose Cytarabine Induction Followed by Consolidation of Clofarabine Plus Low-Dose Cytarabine Alternating With Decitabine in Frontline Acute Myeloid Leukemia (AML) and High-Risk Myelodysplastic Syndrome (MDS)
Brief Title: Clofarabine Plus Low-Dose Cytarabine Induction and Decitabine Consolidation in Frontline Acute Myeloid Leukemia (AML) and High-Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eisai Inc. (Industry); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0039; NCI-2012-01622 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-10-21; First posted 2008-10-23 (Estimated); Results first posted 2016-02-26 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-06

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndrome; AML; MDS; Clofarabine; Ara-C; Cytarabine; Decitabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Clofarabine; Cytarabine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clofarabine + Cytarabine + Decitabine (Experimental): Clofarabine 20 mg/m^2 by vein (IV) as a 1- to 2-hour intravenous infusion daily for 5 days. Cytarabine 20 mg subcutaneously twice daily for 10 days, administered 3 to 6 hours following the start of the clofarabine infusions. Decitabine 20 mg/m^2 as a 1- to 2-hour infusion daily for 5 days.
  Interventions: Drug: Clofarabine; Drug: Cytarabine; Drug: Decitabine

INTERVENTIONS:
Drug: Clofarabine — 20 mg/m^2 by vein as a 1- to 2-hour intravenous infusion daily for 5 days.
  Other Names: Clolar®; Clorarex
Drug: Cytarabine — 20 mg subcutaneously twice daily for 10 days, administered 3 to 6 hours following the start of the clofarabine infusions.
  Other Names: Cytosar-U®; Ara-C; Arabinosylcytosine
Drug: Decitabine — 20 mg/m^2 as a 1- to 2-hour infusion daily for 5 days.
  Other Names: Dacogen®

SUMMARY:
The goal of this clinical research study is to learn if clofarabine given in combination with cytarabine and decitabine can help to control the disease in patients with AML or MDS who are 60 years old or older. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Clofarabine is designed to interfere with the growth and development of cancer cells.

Cytarabine is designed to insert itself into DNA (the genetic material of cells) of cancer cells and stop the DNA from repairing itself.

Decitabine is designed to damage the DNA of cells, which may cause cancer cells to die.

Study Drug Administration:

If you are found eligible to take part in this study, on Days 1-5, you will receive clofarabine through a needle in your vein over 1-2 hours.

On Days 1-10, you will receive cytarabine by injection twice a day.

You may receive up to 2 cycles at this dose and schedule. There are 10 days in each cycle.

Consolidation Cycles:

If you show a response to the treatment, you can then continue with up to a total of 17 more cycles of therapy, which will be called "consolidation cycles". Not every participant may be able to receive all 17 consolidation cycles. The actual number that you will receive depends on whether or not you maintain the response and how you are able to tolerate ongoing therapy. There will be 4-7 weeks in between each consolidation cycle depending on any side effects you may be having and your blood counts.

For consolidation cycles 1, 2, 6, 7, 8, 12, 13, and 14, you will receive clofarabine and cytarabine, but the schedule will be different. On Days 1-3 you will receive clofarabine by vein. On Days 1-7, you will receive cytarabine by vein. On the days when you receive both clofarabine and cytarabine (Days 1-3), the clofarabine will be given about 3-6 hours before the cytarabine injections. You can be taught to give cytarabine injections to yourself. In this case, you can leave the clinic after receiving clofarabine. You will be required to record the injections of cytarabine in a diary unless you receive the treatments while you are in the hospital.

During consolidation cycles 3-5, 9-11, and 15-17, you will receive decitabine only. Decitabine will be given through a needle in your vein over 1-2 hours on Days 1-5. During the decitabine cycles, you may be treated at home, but must return to MD Anderson for study visits before the start of each cycle.

If you do not achieve a response after the first 2 cycles of treatment with clofarabine and cytarabine, you can stay on study and receive 3 cycles of decitabine alone (same dose and schedule as the consolidation course). If you achieve a response after the 3 decitabine cycles, you can continue with the consolidation cycles. If there is no evidence of response after the 3 decitabine cycles, you may be taken off study.

Study Visits:

On Day 1 of every cycle, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will have a performance status evaluation.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.

About 3 weeks after your first course, you may have a bone marrow aspirate to check the status of the disease. To collect a bone marrow aspirate, an area of the hip is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle. After that, you will have a bone marrow aspirate every 2 weeks (or more often if your doctor feels it is necessary). If your routine blood tests indicate that there is still leukemia, you may not need to have the bone marrow samples collected.

You will need to stay in Houston for up to the first 5 weeks of treatment. After that, you will need to return to Houston before each cycle and to receive the clofarabine treatments. Decitabine-only consolidation cycles can be given by your local oncologist. In either case, you can have check-up visits and blood tests with your local doctor between treatments.

Length of Study:

You can stay on study for up to 19 cycles. You will be taken off study early if you experience any intolerable side effects. You may be taken off study early if the disease gets worse.

Follow-up Visits:

Once you are off active treatment but as long as you are still part of the study, every 3-6 months you will have blood (1 tablespoon) drawn to check the status of the disease and your overall health.

This is an investigational study. Clofarabine is FDA approved and commercially available for use in pediatric patients with ALL. Its use in patients with AML is experimental.

Cytarabine is FDA approved and commercially available for use in patients with AML.

Decitabine is FDA approved and commercially available for use in patients with MDS, but its use for patients with AML is investigational.

Up to 120 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated AML and high-risk MDS (>/= 10% blasts or >/= IPSS intermediate-2). Prior therapy with hydroxyurea, biological or targeted therapy (e.g. flt3 inhibitors, other kinase inhibitors, azacitidine), or hematopoietic growth factors is allowed.
2. Age >/= 60 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
4. Adequate hepatic (serum total bilirubin </= 1.5 x ULN, serum glutamate pyruvate transaminase (SGPT) and/or serum glutamate oxaloacetate transaminase (SGOT) </= 2.5 x ULN) and renal function (creatinine </= 1.5 mg/dL).
5. Sign written informed consent

Exclusion Criteria:

1. Cardiac ejection fraction < 40%.
2. Prior therapy with clofarabine or decitabine.
3. Active and uncontrolled disease/infection as judged by the treating physician.
4. Pregnancy
5. Acute promyelocytic leukemia (APL).
6. Women of childbearing potential and men who do not practice contraception.
7. Women of childbearing potential and men must agree to use contraception prior to study entry and for the duration of study participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2008-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 20, 2008 through October 24, 2011. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Clofarabine + Cytarabine + Decitabine: Clofarabine 20 mg/m^2 by vein (IV) as 1-2 hour intravenous infusion daily for 5 days; Cytarabine 20 mg subcutaneously twice daily for 10 days, administered 3-6 hours following start of clofarabine infusions; Decitabine 20 mg/m^2 as 1-2 hour infusion daily for 5 days.
Period: Overall Study
Arm/Group | Clofarabine + Cytarabine + Decitabine
Started | 122
Completed | 119
Not Completed | 3
Not completed — Ineligible | 3

BASELINE CHARACTERISTICS:
Groups:
- Clofarabine + Cytarabine + Decitabine: Clofarabine 20 mg/m^2 IV as 1-2 hour intravenous infusion daily for 5 days; Cytarabine 20 mg subcutaneously twice daily for 10 days, administered 3-6 hours following start of clofarabine infusions; Decitabine 20 mg/m^2 as 1-2 hour infusion daily for 5 days.
Arm/Group | Clofarabine + Cytarabine + Decitabine
Number analyzed (Participants) | 122
Age, Continuous [Median (Full Range); unit: years] | 68 [60 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 78
Region of Enrollment [Number; unit: participants]
  United States | 122

OUTCOME MEASURES:

1. Primary Outcome: Disease-free (DFS) or Relapse-free Survival (RFS) Time
Description: Disease (DFS) or Relapse-free survival (RFS): Time from date of treatment start until the date of first objective documentation of disease-relapse; Bone marrow aspirate and/or biopsy starting on day 21 (+/- 7 days) of therapy and then every 2 weeks (+/- 7 days) as required by leukemia evolution until remission or non-response. Among participants who achieved CR or CRp, RFS was defined as the time interval between the date of response (ie CR or CRp) and the date of relapse or date of death, whichever occurs first. CR or CRp participants who were alive and relapse-free were censored at the off-study date. Full range reflects time to disease progression only, therefore does not reflect a lesser survival time due to other reasons than disease progression/relapse.
Time Frame: Evaluated from treatment date until date of disease progression/relapse, followed for 5 years/60 months.
Population: One participant of 119 treated was not evaluable for outcome.
Measure: Median (Full Range); unit: Months
Arm/Group | Clofarabine + Cytarabine + Decitabine
Number analyzed (Participants) | 118
Months | 15.9 [0.3 to 48.3]

2. Primary Outcome: Complete Remission (CR) Rate for First 60 Participants
Description: All responses were defined as per IWG criteria (2003) where CR Rate defined as number of participants with CR out of total treated participants. Complete remission (CR): Disappearance of all clinical and/or radiologic evidence of disease. Neutrophil count > 1.0 times 10^9/L and platelet count > 100 times 10^9/L, and normal bone marrow differential (< 5% blasts). Bone marrow aspirate and/or biopsy starting on day 21 (+/- 7 days) of therapy.
Time Frame: Evaluation following two 10 day cycles on day 21 of therapy, continuing up to 210 days
Population: The outcome population consisted of first sixty participants enrolled between October 2008 and January 2010, of whom 59 were evaluable for response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Clofarabine + Cytarabine + Decitabine
Number analyzed (Participants) | 59
Percentage of Participants | 58

3. Primary Outcome: Median Overall Survival (OS)
Description: Overall survival (OS): Time from date of treatment start until date of death due to any cause.
Time Frame: Evaluated from treatment date until date of death, followed for 5 years/60 months.
Population: One participant of 119 treated was not evaluable for outcome.
Measure: Median (Full Range); unit: Months
Arm/Group | Clofarabine + Cytarabine + Decitabine
Number analyzed (Participants) | 118
Months
  Overall Survival | 11.1 [0.2 to 53.9]
  Overall Survival among Responders ((n=86) | 21.1 [1.3 to 53.9]

4. Primary Outcome: Number of Participants With Complete Remission [Complete Response (CR), Complete Response With Platelet Recover (CRp) or Complete Response With Incomplete Marrow Recovery (CRi)]
Description: All responses were defined as per IWG criteria (2003) where CR Rate defined as number of participants with CR out of total treated participants. Complete remission (CR): Disappearance of all clinical and/or radiologic evidence of disease. Neutrophil count > 1.0 times 10^9/L and platelet count > 100 times 10^9/L, and normal bone marrow differential (< 5% blasts). Complete response with incomplete marrow recovery (CRi), defined as CR above, but without normal blood counts. Bone marrow aspirate and/or biopsy starting on day 21 (+/- 7 days) of therapy.
Time Frame: Beginning assessment following two 10-day induction cycles through an additional re-induction cycle, up to 40 days
Population: One participant of 119 treated was not evaluable for response. Twenty-two participants required re-induction.
Measure: Number; unit: Participants
Groups:
- Induction Clofarabine + Cytarabine + Decitabine; Re-Induction: Clofarabine 20 mg/m^2 IV as 1-2 hour intravenous infusion daily for 5 days; Cytarabine 20 mg subcutaneously twice daily for 10 days, administered 3-6 hours following start of clofarabine infusions; Decitabine 20 mg/m^2 as 1-2 hour infusion daily for 5 days.
Arm/Group | Induction Clofarabine + Cytarabine + Decitabine | Re-Induction
Number analyzed (Participants) | 118 | 22
Participants
  CR | 60 | 12
  CRp/CRi | 9 | 4

5. Secondary Outcome: Event Free Survival (EFS)
Description: EFS is defined as length of time after primary treatment for a cancer ends that the participant remains free of certain complications or events that the treatment was intended to prevent or delay, for example but not exclusive of hematologic and non-hematologic toxicities, cumulative toxicities with consolidation courses, or emergence of resistance to the chemotherapy component of treatment.
Time Frame: Follow up up to 5 years/60 months.
Population: Of 119 enrolled, one participant was not evaluable for response.
Measure: Median (Full Range); unit: Months
Arm/Group | Clofarabine + Cytarabine + Decitabine
Number analyzed (Participants) | 118
Months | 7.7 [0.2 to 49.5]

6. Secondary Outcome: Overall Response Rate (CR, CRp/CRi and PR)
Description: IWG Response criteria (2003): Complete remission (CR): Disappearance of all clinical and/or radiologic evidence of disease. Neutrophil count > 1.0 times 10^9/L and platelet count > 100 times 10^9/L, and normal bone marrow differential (< 5% blasts). Complete Remission without Platelet Recovery (CRp): Peripheral blood and bone marrow results as for CR, but with platelet counts of < 100 x 10^9/L or Complete remission with incomplete marrow recovery (CRi), defined as CR above, but without normal blood counts; Partial Remission (PR): Blood count recovery as for CR, but with both a decrease in marrow blasts of at least 50% and not more than 6 to 25% abnormal cells in the marrow. Participants not achieving a complete remission following first induction course, can receive a second induction course at least 28 days following first to optimize response if possible.
Time Frame: Beginning assessment following two 10-day induction cycles through an additional re-induction cycle, up to 40 days
Population: Of 119 enrolled, one participant was not evaluable for response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Clofarabine + Cytarabine + Decitabine
Number analyzed (Participants) | 118
Percentage of Participants | 73

ADVERSE EVENTS:
Time Frame: Adverse events captured from the time of the first treatment, until 30 days after the last dose of drug. Treatment could last up to nineteen 10-day cycles (approximately 200 days).
Arm/Group | Clofarabine + Cytarabine + Decitabine
Serious Adverse Events (participants affected / at risk) | 12/119
Other Adverse Events (participants affected / at risk) | 67/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine + Cytarabine + Decitabine (N=119)
Sudden death (General disorders) | 2 (2)
Death (General disorders) | 2 (2)
Infection (Infections and infestations) | 5 (5) — Infection secondary to myelosuppression
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 7 — Myelosuppression
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine + Cytarabine + Decitabine (N=119)
Abdominal infection (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3)
Allergic rhinitis (Immune system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Bilirubin increased (Investigations) | 4 (4)
Blood/Bone Marrow (Other) (Blood and lymphatic system disorders) | 2 (2)
Cardiac arrhythmia (Other) (Cardiac disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Constipation (Psychiatric disorders) | 2 (2)
Creatinine increased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 31 (43)
Fever (General disorders) | 7 (7)
Headache (Nervous system disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Hemorrhage/Bleeding (Other) (Blood and lymphatic system disorders) | 3 (3)
Hypersensitivity (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Infection (Infections and infestations) | 26 (40)
Infection - Neck (Infections and infestations) | 1 (1)
Infection (Other) - 10021789 / CTCAE3.M10 (Infections and infestations) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Neurology (Other) (Nervous system disorders) | 1 (1)
Pain (Other) (General disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary (Other) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3)
Renal failure (Renal and urinary disorders) | 6 (6)
Seizure (Nervous system disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes